CLINICAL TRIAL: NCT02454127
Title: Effectiveness of Four Dietary Treatment Strategies for Metabolic Syndrome: a Prospective Randomized Trial
Brief Title: Effectiveness of Four Popular Diet Strategies for Weight Loss and Cardiac Risk Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DANS0001
Record Dates: First submitted 2015-05-20; First posted 2015-05-27 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; Cardiovascular Disease; Metabolic Syndrome
Keywords: nutrition; popular diets; weight loss; lifestyle; counseling
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Metabolic Syndrome; Weight Loss | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atkins Diet (Active Comparator): Atkins Diet (dietary counseling)
  Interventions: Behavioral: Atkins Diet
- Zone Diet (Active Comparator): Zone Diet (dietary counseling)
  Interventions: Behavioral: Zone Diet
- Weight Watchers Diet (Active Comparator): Weight Watchers Diet (dietary counseling)
  Interventions: Behavioral: Weight Watchers Diet
- Ornish Diet (Active Comparator): Ornish Diet (dietary counseling)
  Interventions: Behavioral: Ornish Diet

INTERVENTIONS:
Behavioral: Atkins Diet — Dietary counseling for 1 year
  Arms: Atkins Diet
Behavioral: Zone Diet — Dietary counseling for 1 year
  Arms: Zone Diet
Behavioral: Weight Watchers Diet — Dietary counseling for 1 year
  Arms: Weight Watchers Diet
Behavioral: Ornish Diet — Dietary counseling for 1 year
  Arms: Ornish Diet

SUMMARY:
A single-center randomized trial at an academic medical center in Boston, Mass, of overweight or obese adults with known hypertension, dyslipidemia, or fasting hyperglycemia. Participants were enrolled starting July 18, 2000, and randomized to 4 popular diet groups until January 24, 2002.

DETAILED DESCRIPTION:
Objective: To assess adherence rates and the effectiveness of 4 popular diets (Atkins, Zone, Weight Watchers, and Ornish) for weight loss and cardiac risk factor reduction.

Design, Setting, and Participants: A single-center randomized trial at an academic medical center in Boston, Mass, of overweight or obese adults with known hypertension, dyslipidemia, or fasting hyperglycemia. Participants were enrolled starting July 18, 2000, and randomized to 4 popular diet groups until January 24, 2002.

Intervention: A total of 160 participants were randomly assigned to either Atkins (carbohydrate restriction, n=40), Zone (macronutrient balance, n=40), Weight Watchers (calorie restriction, n=40), or Ornish (fat restriction, n=40) diet groups. After 2 months of maximum effort, participants selected their own levels of dietary adherence.

Main Outcome Measures: One-year changes in baseline weight and cardiac risk factors, and self-selected dietary adherence rates per self-report. Outcome measures included body weight, total cholesterol, LDL-C, HDL-C, triglycerides, hsCRP, insulin, glucose.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-42;
* At least one metabolic cardiac risk factor

Exclusion Criteria:

* Age under 18 years;
* Insulin therapy;
* Unstable chronic illness;
* Unwilling to follow dietary advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2000-07; Primary Completion 2003-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Dansinger, MD, Principal Investigator — Tufts Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Peer-reviewed publication

REFERENCES:
- [Result] Dansinger ML, Gleason JA, Griffith JL, Selker HP, Schaefer EJ. Comparison of the Atkins, Ornish, Weight Watchers, and Zone diets for weight loss and heart disease risk reduction: a randomized trial. JAMA. 2005 Jan 5;293(1):43-53. doi: 10.1001/jama.293.1.43. PMID 15632335

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Started | 40 | 40 | 40 | 40
Completed | 21 | 26 | 26 | 20
Not Completed | 19 | 14 | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) | 51 (9) | 49 (10) | 49 (12) | 49 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 23 | 17 | 81
  Male | 19 | 20 | 17 | 23 | 79
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 40 | 160

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Change from baseline body weight at 1 year, measured in kilograms
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
kg | -2.1 (4.8) | -3.2 (6.0) | -3.0 (4.9) | -3.3 (7.3)

2. Secondary Outcome: Total Cholesterol
Description: Change in total cholesterol from baseline at 1 year, measured in mg/dL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline data.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dL | -4.3 (23) | -10.1 (35) | -8.2 (24) | -10.8 (21)

3. Secondary Outcome: LDL Cholesterol
Description: Change from baseline LDL cholesterol at 1 year, measured in mg/dL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dL | -7.1 (24) | -11.8 (34) | -9.3 (27) | -12.6 (19)

4. Secondary Outcome: HDL Cholesterol
Description: Change from baseline HDL cholesterol at 1 year, measured in mg/dL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dL | 3.4 (7.1) | 3.3 (10.3) | 3.4 (9.9) | -0.5 (6.5)

5. Secondary Outcome: Triglycerides
Description: Change from baseline triglycerides at 1 year, measured in mg/dL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dL | -1.2 (84) | 2.5 (147) | -12.7 (61) | 5.6 (36)

6. Secondary Outcome: Glucose
Description: Change from baseline glucose at 1 year, measured in mg/dL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/dL | 1.4 (30) | -4.2 (18) | -4.7 (19) | -4.1 (30)

7. Secondary Outcome: Insulin
Description: Change from baseline insulin at 1 year, measured in microIU/mL
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values
Measure: Mean (Standard Deviation); unit: microIU/ml
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
microIU/ml | -1.2 (6.7) | -5.4 (14) | -2.6 (6.1) | -3.0 (6.3)

8. Secondary Outcome: C-reactive Protein
Description: Change from baseline high-sensitivity CRP at 1 year, measured in mg/L
Time Frame: 1 year
Population: Intent-to-treat analysis. Missing data were replaced with baseline values.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Number analyzed (Participants) | 40 | 40 | 40 | 40
mg/L | -0.70 (2.1) | -0.58 (2.1) | -0.58 (1.3) | -0.88 (2.4)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Clinically significant adverse events likely related to dietary adherence
Arm/Group | Atkins Diet | Zone Diet | Weight Watchers Diet | Ornish Diet
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The protocol provided dietary advice rather than food. The attrition rate was 35% to 50% in each group. Missing data were replaced with baseline data for intent-to-treat analysis. Long-term safety beyond 1-year was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes